CLINICAL TRIAL: NCT01032395
Title: A Phase 3, Randomized, Controlled, Open Label Study to Evaluate the Immunogenicity, Safety, and Tolerability of MF59-Adjuvanted Versus Non-Adjuvanted Vaccines Against Novel H1N1 Virus in Patients With Chronic Pulmonary Disease, Chronic Heart Disease, or Diabetes Mellitus
Brief Title: Immunogenicity, Safety, and Tolerability of an MF59-Adjuvanted Versus Non-Adjuvanted Influenza Vaccines in Patients With Chronic Pulmonary Disease, Chronic Heart Disease, or Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiltern Pesquisa Clinica Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V111_16TP
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: H1N1 Influenza Virus; Chronic Pulmonary Disease; Chronic Heart Disease; Diabetes Mellitus
Keywords: H1N1; Pulmonary Disease; Heart Disease; Diabetes; Influenza; immunogenicity; safety; tolerability
MeSH Terms: conditions — Diabetes Mellitus; Lung Diseases; Heart Diseases; Influenza, Human | interventions — focetria; fluad vaccine

ARMS (4):
- Chronic Disease Subjects Receiving Vaccine with Adjuvant (Experimental): Each subject received two doses of vaccine with adjuvant (Focetria® or Fluad®), the first on Study Day 1, and the second on Study Day 22.
  Interventions: Biological: Focetria®; Biological: Fluad®
- Chronic Disease Subjects Receiving Vaccine without Adjuvant (Experimental): Each subject received two doses of vaccine without adjuvant (Begrivac®), the first on Study Day 1, and the second on Study Day 22.
  Interventions: Biological: Begrivac®
- Healthy Subjects Receiving Vaccine with Adjuvant (Experimental): Each subject received two doses of vaccine with adjuvant (Focetria® or Flaud®), the first on Study Day 1, and the second on Study Day 22.
  Interventions: Biological: Focetria®; Biological: Fluad®
- Healthy Subjects Receiving Vaccine without Adjuvant (Experimental): Each subject received two doses of vaccine without adjuvant (Begrivac®), the first on Study Day 1, and the second on Study Day 22.
  Interventions: Biological: Begrivac®

INTERVENTIONS:
Biological: Focetria® — 7.5 ug of HA antigen; adjuvanted; monovalent
  Arms: Chronic Disease Subjects Receiving Vaccine with Adjuvant; Healthy Subjects Receiving Vaccine with Adjuvant
Biological: Fluad® — 15 ug of HA antigen; adjuvanted; trivalent
  Arms: Chronic Disease Subjects Receiving Vaccine with Adjuvant; Healthy Subjects Receiving Vaccine with Adjuvant
Biological: Begrivac® — 15 ug of antigen; non-adjuvanted; trivalent
  Arms: Chronic Disease Subjects Receiving Vaccine without Adjuvant; Healthy Subjects Receiving Vaccine without Adjuvant

SUMMARY:
This is a phase III, randomized, controlled, open label study with two vaccine regimens. The study will assess the relative safety and immunogenicity of vaccine regimens comparing adjuvanted versus non-adjuvanted formulations of A(H1N1) inactivated influenza virus vaccine in subjects with Chronic Pulmonary Disease, Chronic Heart Disease, or Diabetes Mellitus, and to compare safety and immunogenicity data with a contemporaneously enrolled control group of age-comparable, healthy subjects.

Because certain individuals may be hypo-responsive to influenza vaccination, additional studies with high-risk groups are warranted in order to determine the optimal vaccine formulation and dosing schedule for prevention of novel H1N1 virus infection.

ELIGIBILITY:
Inclusion Criteria:

For Subjects with Chronic Diseases:

* Subjects between 18 and 70 years of age (inclusive)
* Any sex or ethnicity
* Outpatient or hospitalized subjects
* Confirmed diagnosis of chronic pulmonary and/or cardiac, and/or diabetes mellitus based on the investigator's assessment (subjects may present one or more of such conditions)
* Childbearing potential women must be willing to use an acceptable contraceptive method. Acceptable contraceptive methods are defined as one or more of the following:

  1. Hormone contraceptive (such as oral, injectable, transdermal patch, subcutaneous implant, cervical ring)
  2. Barrier (condom with spermicide or diaphragm with spermicide) at each intercourse and during the whole intercourse
  3. Intra-uterine device (IUD)
  4. Monogamous relation with vasectomized partner (must have been vasectomized at least six months before the volunteer entered the study)
* Subjects capable of following all the study procedures and available for all visits scheduled to the investigation site
* Subjects capable of understanding the nature and risk of the study proposed and sign the consent form
* The study subjects may have other underlying chronic diseases that do not involve immunosuppression (e.g. osteoarticular diseases, stable, non-progressive, non-severe neurologic disorders without cognitive impairment, ophthalmologic diseases, hypothyroidism, etc.), but their symptoms/signs must be under control through medical follow-ups and drug therapy

For Healthy Subjects:

* Subjects between 18 and 70 years of age (inclusive)
* Any sex and ethnicity
* Subjects with good health as determined by medical history, physical evaluation, and investigator's clinical opinion
* Childbearing potential women must be willing to use an acceptable contraceptive method. Acceptable contraceptive methods are defined as one or more of the following:

  1. Hormone contraceptive (such as oral, injectable, transdermal patch, subcutaneous implant, cervical ring)
  2. Barrier (condom with spermicide or diaphragm with spermicide) at each intercourse and during the whole sexual intercourse
  3. Intra-uterine device (IUD)
  4. Monogamous relation with vasectomized partner (must have been vasectomized for at least six months before the volunteer entered the study)
* Subjects capable of respecting all the study procedures and available for all the visits scheduled at the investigation site
* Subjects capable of understanding the nature and risk of the study proposed and sign the consent form

Exclusion Criteria:

For Subjects with Chronic Diseases

* Previous laboratory confirmed diagnosis of an infection by the novel H1N1 virus
* Administration of other vaccine against the novel H1N1 virus within 3 months prior to inclusion in the study
* Any recent vaccine given within the last 21 days (inclusive)
* History of allergic reaction to an influenza vaccine in the past, or a current or previous occurrence of allergy to egg or egg protein, kanamycin, and neomycin sulfate
* Acute febrile disease (vaccination may be delayed up to 3 days after the resolution of the symptoms)
* History of cancer, except for skin cancer, including Kaposi's Sarcoma, basal cell carcinoma, and non-invasive malignancy related to HPV
* History of chronic hepatic or renal disease
* History of cognitive disorders
* History of progressive or severe neurological disorders, including Guillain-Barré Syndrome
* Pregnancy or breast-feeding
* Use of immunomodulatory therapy, including cyclosporin,interleukins, and interferons, within 3 months prior to inclusion in the study
* Receipt of parenteral immunoglobulin, hemotherapy, and/or plasma derivatives within 3 months prior to inclusion in the study
* Life expectancy of at least 12 months
* Receipt of any investigational product within 12 months prior to inclusion in the study

For Healthy Subjects:

* Previous laboratory confirmed diagnosis of an infection by the new virus H1N1
* Receipt of another vaccine against the new virus H1N1 within 3 months prior to inclusion in the study
* Any recent vaccine given within the last 21 days (inclusive)
* History of allergic reaction to influenza vaccine in the past, or a current or previous allergy to egg or egg protein, kanamycin, and neomycin sulfate
* Acute febrile disease (the vaccination may be delayed up to 3 days after symptoms resolution)
* Pregnancy or breast-feeding
* Receipt of parenteral immunoglobulin, hemotherapy, and/or plasma derivatives within 3 months prior to inclusion in the study
* Receipt of any investigational product within 12 months prior to inclusion in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Geometric Mean HI Titer by Visit | 13 months after vaccination (Day 1, Day 22, Day 43, Day 133, Day 223 and Day 403)
  Geometric mean hemagglutinin inhibition (HI) titer = GMT
Geometric Mean Ratio by Visit | 13 months after vaccination (Day 22/Day1, Day 43/Day 1, Day 43/Day 22, Day 133/Day 43, Day 223/Day 43 and Day 403/Day 223)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with chronic diseases (chronic cardiac diseases, chronic pulmonary diseases and diabetes mellitus).
Ratio of Immunogenicity Data by Visit (Vaccine With Adjuvant : Vaccine Without Adjuvant) | 13 months after vaccination (Day 1, Day 22, Day 22/Day1, Day 43, Day 43/Day 1, Day 43/Day 22, Day 133, Day 133/Day 43, Day 223, Day 223/Day 43 and Day 403, Day 403/Day 223)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with chronic diseases (chronic cardiac diseases, chronic pulmonary diseases and diabetes mellitus). Comparisons were made by vaccine group using ratios of immunogenicity data and were presented with 95% confidence intervals.
Percentage of Subjects Who Reached Seroprotection by Visit | 13 months after vaccination (Day 22, Day 43, Day 133, Day 223 and Day 403)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with chronic diseases (chronic cardiac diseases, chronic pulmonary diseases and diabetes mellitus). The percentage of subjects that reached seroprotection in comparison to the pre-vaccination result are presented by visit. Seroprotection was defined as HI titer ≥40.
Percent of Subjects Who Seroconverted or Had a Significant Increase in Geometric Mean Titer by Visit | 13 Months after vaccination (Day 22, Day 43, Day 133, Day 223 and Day 403)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with chronic diseases (chronic cardiac diseases, chronic pulmonary diseases and diabetes mellitus). The percentage of subjects that reached seroconversion or had a significant increase in comparison to the pre-vaccination result were presented by visit. Seroconversion or a significant increase was defined as HI titer ≥40 in subjects with negative results at pre-vaccination (HI titer <10) or an increase of at least 4 times in HI titer for individuals with positive results at pre-vaccination (HI titer >10) at Day 22 and Day 43 in comparison to the pre-vaccination result.
Difference in the Seroprotection Rates by Visit (Vaccine With Adjuvant - Vaccine Without Adjuvant) | 13 Months after vaccination (Day 22, Day 43, Day 133, Day 223 and Day 403)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with chronic diseases (chronic cardiac diseases, chronic pulmonary diseases and diabetes mellitus). Comparisons were made by vaccine group using differences in the percentage of subjects with seroprotection and were presented with 95% confidence intervals.
Differences in the Seroconversion Rates or Significant Increase by Visit (Vaccine With Adjuvant - Vaccine Without Adjuvant) | 13 Months after vaccination (Day 22, Day 43, Day 133, Day 223 and Day 403)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with chronic diseases (chronic cardiac diseases, chronic pulmonary diseases and diabetes mellitus). Comparisons were made by vaccine group using differences in the percentage of subjects with seroconversion/significant increase and were presented with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Centro de Estudos de Pneumologia da Faculdade de Medicina do ABC, Santo André, São Paulo
  - Instituto de Ensino e Pesquisa em Geriatria e Gerontologia, São Paulo, São Paulo

REFERENCES:
- [Background] ANZIC Influenza Investigators; Webb SA, Pettila V, Seppelt I, Bellomo R, Bailey M, Cooper DJ, Cretikos M, Davies AR, Finfer S, Harrigan PW, Hart GK, Howe B, Iredell JR, McArthur C, Mitchell I, Morrison S, Nichol AD, Paterson DL, Peake S, Richards B, Stephens D, Turner A, Yung M. Critical care services and 2009 H1N1 influenza in Australia and New Zealand. N Engl J Med. 2009 Nov 12;361(20):1925-34. doi: 10.1056/NEJMoa0908481. Epub 2009 Oct 8. PMID 19815860
- [Background] Bridges CB, Katz JM, Levandowski RA, Cox NJ. Inactivated influenza vaccines. In. Plotkin SA, Orenstein WA, Offit PA. Vaccines 5th ed. WB Saunders. Phila PA 2008; 291-309
- [Background] Clark TW, Pareek M, Hoschler K, Dillon H, Nicholson KG, Groth N, Stephenson I. Trial of 2009 influenza A (H1N1) monovalent MF59-adjuvanted vaccine. N Engl J Med. 2009 Dec 17;361(25):2424-35. doi: 10.1056/NEJMoa0907650. Epub 2009 Sep 10. PMID 19745215
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] Dominguez-Cherit G, Lapinsky SE, Macias AE, Pinto R, Espinosa-Perez L, de la Torre A, Poblano-Morales M, Baltazar-Torres JA, Bautista E, Martinez A, Martinez MA, Rivero E, Valdez R, Ruiz-Palacios G, Hernandez M, Stewart TE, Fowler RA. Critically Ill patients with 2009 influenza A(H1N1) in Mexico. JAMA. 2009 Nov 4;302(17):1880-7. doi: 10.1001/jama.2009.1536. Epub 2009 Oct 12. PMID 19822626
- [Background] Jain S, Kamimoto L, Bramley AM, Schmitz AM, Benoit SR, Louie J, Sugerman DE, Druckenmiller JK, Ritger KA, Chugh R, Jasuja S, Deutscher M, Chen S, Walker JD, Duchin JS, Lett S, Soliva S, Wells EV, Swerdlow D, Uyeki TM, Fiore AE, Olsen SJ, Fry AM, Bridges CB, Finelli L; 2009 Pandemic Influenza A (H1N1) Virus Hospitalizations Investigation Team. Hospitalized patients with 2009 H1N1 influenza in the United States, April-June 2009. N Engl J Med. 2009 Nov 12;361(20):1935-44. doi: 10.1056/NEJMoa0906695. Epub 2009 Oct 8. PMID 19815859
- [Background] Kumar A, Zarychanski R, Pinto R, Cook DJ, Marshall J, Lacroix J, Stelfox T, Bagshaw S, Choong K, Lamontagne F, Turgeon AF, Lapinsky S, Ahern SP, Smith O, Siddiqui F, Jouvet P, Khwaja K, McIntyre L, Menon K, Hutchison J, Hornstein D, Joffe A, Lauzier F, Singh J, Karachi T, Wiebe K, Olafson K, Ramsey C, Sharma S, Dodek P, Meade M, Hall R, Fowler RA; Canadian Critical Care Trials Group H1N1 Collaborative. Critically ill patients with 2009 influenza A(H1N1) infection in Canada. JAMA. 2009 Nov 4;302(17):1872-9. doi: 10.1001/jama.2009.1496. Epub 2009 Oct 12. PMID 19822627
- [Background] Vaillant L, La Ruche G, Tarantola A, Barboza P; epidemic intelligence team at InVS. Epidemiology of fatal cases associated with pandemic H1N1 influenza 2009. Euro Surveill. 2009 Aug 20;14(33):19309. doi: 10.2807/ese.14.33.19309-en. PMID 19712643